CLINICAL TRIAL: NCT02441985
Title: rTMS Therapy for Primary Orthostatic Tremor: A Novel Treatment Approach
Brief Title: rTMS Therapy for Primary Orthostatic Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Organization for Rare Disorders (Other); Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201500347
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Primary Orthostatic Tremor
Keywords: Primary orthostatic tremor
MeSH Terms: conditions — Primary orthostatic tremor | interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS Stimulation (Experimental): rTMS will be delivered over each cerebellar hemisphere, using a 70mm figure-of-eight coil connected to a Magstim RapidStim2 machine while positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere. The RMT will be defined as the lowest stimulation intensity required to evoke a 50 μV potential in a target muscle. The inion will be taken as the boundary between the posterior cerebellum and the occipital cortex. Therefore the area stimulated will be caudal to the inion to stimulate the posterior cerebellum.
  Interventions: Device: Magstim RapidStim2; Other: Fullerton Advanced Balance (FAB) Scale; Other: Timed "Up & Go" Test (TUG) test; Other: 10m walk test; Other: Tremor electrophysiology; Other: Cerebellar-brain Inhibition (CBI)
- Sham rTMS Stimulation (Sham Comparator): Patients randomized to receive sham treatment will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using sham Magstim RapidStim2 Placebo which produces discharge noise and vibration similar to the real coil without stimulating the cerebral cortex. However, in addition to obvious coil discharge noise, rTMS also causes electrical stimulation of the scalp. The investigator will simulate this experience by attaching surface electrodes underneath the sham coil and in contact with the scalp. The investigator will use an electromyography to administer electrical shocks to the scalp simultaneous to each simulated rTMS train.
  Interventions: Device: Sham Magstim RapidStim2; Other: Fullerton Advanced Balance (FAB) Scale; Other: Timed "Up & Go" Test (TUG) test; Other: 10m walk test; Other: Tremor electrophysiology; Other: Cerebellar-brain Inhibition (CBI)

INTERVENTIONS:
Device: Magstim RapidStim2 — Application of repetitious transcranial magnetic stimulation (TMS) pulses using Magstim RapidStim2 to a specific brain target at predefined stimulation parameters.
  Arms: Real rTMS Stimulation
Device: Sham Magstim RapidStim2 — Same procedure as real rTMS without stimulating the cerebral cortex.
  Arms: Sham rTMS Stimulation
Other: Fullerton Advanced Balance (FAB) Scale — All participants will receive a clinical assessment of balance ability and fall risk.
Other: Timed "Up & Go" Test (TUG) test — All participants will receive a clinical assessment of basic mobility skills by using the TUG test.
Other: 10m walk test — All participants will receive a clinical assessment of walking speed by using the walk test.
Other: Tremor electrophysiology — All participant tremors will by analyzed using an EMG system
Other: Cerebellar-brain Inhibition (CBI) — All participants will have a measure of the cerebellar-brain inhibition (CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.

SUMMARY:
Primary orthostatic tremor(POT) is a rare progressive functionally disabling tremor disorder. The characteristic features of POT are symptoms of unsteadiness in legs reported by patients when they are standing and improvement of symptoms upon walking and sitting. Due to the limited success of other treatment options there is a clear merit in continuing efforts to explore and investigate novel treatment modalities. Transcranial magnetic stimulation (TMS) is a well-established physiological tool to understand brain function. When repetitious TMS pulses are delivered to a specific target at predefined stimulation parameters, it is referred to as rTMS therapy.The investigators propose a novel approach to investigate the clinical and physiological effects of low frequency rTMS therapy in POT. The overarching hypothesis of this study is that low frequency rTMS therapy delivered to the cerebellum will modulate the cerebellar excitability and result in clinical improvements.In order to determine the physiological effects related to rTMS, the tremor physiology will also be recorded with surface electromyography (EMG). The investigator will also record the changes in cerebellum excitability in response to rTMS using cerebello-cortical inhibition (CBI), a well-established TMS parameter.

DETAILED DESCRIPTION:
POT tremors recorded on surface electromyography (EMG) reveal distinct high frequency bursts of 13-18 Hz tremors in the leg muscles. POT was first described in 1984 at the University of Florida. Since then several clinical descriptions have been published however despite this knowledge for thirty years, treatment opportunities for POT have remained poor. Several medications have been tried, but the results have been disappointing. Thalamic deep brain stimulation (DBS) surgery, which is an invasive therapy approved by the FDA for treatment of essential tremor, was recently investigated in POT but the early results have only been partially successful. In clinical descriptions, POT has been observed to be associated with clinical features of cerebellar dysfunction such as dysmetria and gait ataxia. Positron emission tomography (PET) imaging has shown an increased activation of bilateral cerebellum related either to a mismatch between the peripheral afferent and the cerebellar efferent traffic or to a primary disorder of the cerebellum. MRI study has confirmed a cerebellar atrophy in POT and finally transcranial magnetic stimulation (TMS), has shown POT can be reset by stimulation of the cerebellum. The primary goal of this study is to test the efficacy of low frequency rTMS therapy in POT. The first aim of the study is to determine the clinical impact of 1-Hz rTMS therapy in POT when delivered to the cerebellum. This impact will be evaluated by the clinical scoring of leg tremors in standing posture, and the functional assessment of gait mobility. The second aim of this study is to determine the physiological effects of 1-Hz rTMS therapy in POT when delivered to the cerebellum. The investigator will determine the effects on the amplitude and frequency of tremors recorded with surface EMG. They will also determine the effects on the cerebello-cortical inhibition measured with TMS. Comparisons will be drawn between before rTMS therapy, immediately or +5 minutes after and 60+ minutes after assessments to determine the time course of effects. In this application, subjects with POT will be enrolled based on clinical history, physical exam and a 13-18 Hz tremor recorded on the surface EMG in accordance with the Consensus Statement of the Movement Disorder Society. Data will be presented as mean (SD) unless otherwise indicated. For each of the outcome variables, the statistical analyst will conduct a mixed model analysis using time and stimulation arm as repeated factors adjusted for baseline values, and subjects as the random factor.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be diagnosed with Primary orthostatic tremor (POT) and be recruited through IRB approved database maintained by the Movement Disorders Center

Exclusion Criteria:

* Pregnancy
* Active seizure disorder
* Significant cognitive impairment
* Presence of a metallic body such as pacemaker, implants, prosthesis,artificial limb or joint, shunt, metal rods and hearing aid

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle-Shukla, M.D., Principal Investigator — Center for Movement Disorders and Neurorestoration
Locations (1):
- Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

REFERENCES:
- [Background] Wagle Shukla A, Vaillancourt DE. Treatment and physiology in Parkinson's disease and dystonia: using transcranial magnetic stimulation to uncover the mechanisms of action. Curr Neurol Neurosci Rep. 2014 Jun;14(6):449. doi: 10.1007/s11910-014-0449-5. PMID 24771105
- [Background] Udupa K, Chen R. Motor cortical plasticity in Parkinson's disease. Front Neurol. 2013 Sep 4;4:128. doi: 10.3389/fneur.2013.00128. PMID 24027555
- [Background] Ugawa Y, Uesaka Y, Terao Y, Hanajima R, Kanazawa I. Magnetic stimulation over the cerebellum in humans. Ann Neurol. 1995 Jun;37(6):703-13. doi: 10.1002/ana.410370603. PMID 7778843
- [Background] Stacy MA, Elble RJ, Ondo WG, Wu SC, Hulihan J; TRS study group. Assessment of interrater and intrarater reliability of the Fahn-Tolosa-Marin Tremor Rating Scale in essential tremor. Mov Disord. 2007 Apr 30;22(6):833-8. doi: 10.1002/mds.21412. PMID 17343274
- [Background] Mathias S, Nayak US, Isaacs B. Balance in elderly patients: the "get-up and go" test. Arch Phys Med Rehabil. 1986 Jun;67(6):387-9. PMID 3487300
- [Background] Ugawa Y, Terao Y, Hanajima R, Sakai K, Furubayashi T, Machii K, Kanazawa I. Magnetic stimulation over the cerebellum in patients with ataxia. Electroencephalogr Clin Neurophysiol. 1997 Sep;104(5):453-8. doi: 10.1016/s0168-5597(97)00051-8. PMID 9344082
- [Background] Roth BJ, Saypol JM, Hallett M, Cohen LG. A theoretical calculation of the electric field induced in the cortex during magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1991 Feb;81(1):47-56. doi: 10.1016/0168-5597(91)90103-5. PMID 1705219
- [Background] Amassian VE, Cracco RQ, Maccabee PJ, Cracco JB. Cerebello-frontal cortical projections in humans studied with the magnetic coil. Electroencephalogr Clin Neurophysiol. 1992 Aug;85(4):265-72. doi: 10.1016/0168-5597(92)90115-r. PMID 1380914
- [Background] Cohen LG, Roth BJ, Nilsson J, Dang N, Panizza M, Bandinelli S, Friauf W, Hallett M. Effects of coil design on delivery of focal magnetic stimulation. Technical considerations. Electroencephalogr Clin Neurophysiol. 1990 Apr;75(4):350-7. doi: 10.1016/0013-4694(90)90113-x. PMID 1691084
- [Background] Werhahn KJ, Taylor J, Ridding M, Meyer BU, Rothwell JC. Effect of transcranial magnetic stimulation over the cerebellum on the excitability of human motor cortex. Electroencephalogr Clin Neurophysiol. 1996 Feb;101(1):58-66. doi: 10.1016/0013-4694(95)00213-8. PMID 8625878
- [Background] Hashimoto M, Ohtsuka K. Transcranial magnetic stimulation over the posterior cerebellum during visually guided saccades in man. Brain. 1995 Oct;118 ( Pt 5):1185-93. doi: 10.1093/brain/118.5.1185. PMID 7496779
- [Background] Deuschl G, Lucking CH, Quintern J. [Orthostatic tremor: clinical aspects, pathophysiology and therapy]. EEG EMG Z Elektroenzephalogr Elektromyogr Verwandte Geb. 1987 Mar;18(1):13-9. German. PMID 3106000
- [Background] Heilman KM. Orthostatic tremor. Arch Neurol. 1984 Aug;41(8):880-1. doi: 10.1001/archneur.1984.04050190086020. PMID 6466163
- [Background] Espay AJ, Duker AP, Chen R, Okun MS, Barrett ET, Devoto J, Zeilman P, Gartner M, Burton N, Miranda HA, Mandybur GT, Zesiewicz TA, Foote KD, Revilla FJ. Deep brain stimulation of the ventral intermediate nucleus of the thalamus in medically refractory orthostatic tremor: preliminary observations. Mov Disord. 2008 Dec 15;23(16):2357-62. doi: 10.1002/mds.22271. PMID 18759339
- [Background] Guridi J, Rodriguez-Oroz MC, Arbizu J, Alegre M, Prieto E, Landecho I, Manrique M, Artieda J, Obeso JA. Successful thalamic deep brain stimulation for orthostatic tremor. Mov Disord. 2008 Oct 15;23(13):1808-11. doi: 10.1002/mds.22001. PMID 18671286
- [Background] Benito-Leon J, Rodriguez J. Orthostatic tremor with cerebellar ataxia. J Neurol. 1998 Dec;245(12):815. doi: 10.1007/s004150050294. No abstract available. PMID 9840357
- [Background] Setta F, Jacquy J, Hildebrand J, Manto MU. Orthostatic tremor associated with cerebellar ataxia. J Neurol. 1998 May;245(5):299-302. doi: 10.1007/s004150050222. No abstract available. PMID 9617712
- [Background] Wills AJ, Thompson PD, Findley LJ, Brooks DJ. A positron emission tomography study of primary orthostatic tremor. Neurology. 1996 Mar;46(3):747-52. doi: 10.1212/wnl.46.3.747. PMID 8618676
- [Background] Manto MU, Setta F, Legros B, Jacquy J, Godaux E. Resetting of orthostatic tremor associated with cerebellar cortical atrophy by transcranial magnetic stimulation. Arch Neurol. 1999 Dec;56(12):1497-500. doi: 10.1001/archneur.56.12.1497. PMID 10593305
- [Background] Deuschl G, Bain P, Brin M. Consensus statement of the Movement Disorder Society on Tremor. Ad Hoc Scientific Committee. Mov Disord. 1998;13 Suppl 3:2-23. doi: 10.1002/mds.870131303. PMID 9827589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10/10 participants who expressed interest in research were randomized
Groups:
- Real rTMS Stimulation First, Then Sham rTMS Stimulation: Participants received single 30 minute long session of real rTMS first that included 900 pulses delivered over the cerebellum, there was washout period of one day before they received sham rTMS dose of 900 pulses over the cerebellum
- Sham rTMS Stimulation First, Then Real rTMS Stimulation: Participants received single 30 minute long session of sham rTMS first that included 900 pulses delivered over the cerebellum, there was washout period of one day before they received real rTMS dose of 900 pulses over the cerebellum
Period: First Intervention (30 Min)
Arm/Group | Real rTMS Stimulation First, Then Sham rTMS Stimulation | Sham rTMS Stimulation First, Then Real rTMS Stimulation
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (One Day)
Arm/Group | Real rTMS Stimulation First, Then Sham rTMS Stimulation | Sham rTMS Stimulation First, Then Real rTMS Stimulation
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (30 Min)
Arm/Group | Real rTMS Stimulation First, Then Sham rTMS Stimulation | Sham rTMS Stimulation First, Then Real rTMS Stimulation
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Real rTMS Stimulation First, Then Sham rTMS Stimulation: Participants freceived 900 pulse of real rTMS
- Sham rTMS Stimulation First, Then Real rTMS Stimulation: Participants received 900 pulse of sham rTMS
- Total: Total of all reporting groups
Arm/Group | Real rTMS Stimulation First, Then Sham rTMS Stimulation | Sham rTMS Stimulation First, Then Real rTMS Stimulation | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.3) | 71.3 (8.3) | 71.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease Duration [Mean (Standard Deviation); unit: years] — How long the participant has had the disease, reported in years.
  years | 14.7 (10.7) | 14.7 (10.7) | 14.7 (10.7)
Standing Duration [Mean (Standard Deviation); unit: seconds] — Video-recorded and timed assessment of standing duration.
  seconds | 97 (74) | 97 (74) | 97 (74)
Tremor Frequency [Mean (Standard Deviation); unit: Hz] — Peak tremor frequency in Hz, calculated from a power analysis of EMG signal of the dominant hand muscle.
  Hz | 15.5 (0.7) | 15.5 (0.7) | 15.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fullerton Advanced Balance (FAB) Scale Total Score After rTMS
Description: The Fullerton Advanced Balance (FAB) Scale is a clinical assessment of balance ability and fall risk. Participants complete 10 physical activity challenges while observed, and their performance is rated on a 0-4 scale, where a higher score a greater ability to balance. Each item is then summed to generate a Total Score, ranging from 0-40, where a higher total score indicates greater overall balance and lower likelihood of fall risk. The reported measure is the change in the FAB Total Score from before and after, where a positive value implies improvement in balance, a negative value indicates a worsening of balance, and 0 indicates no change.
Time Frame: Pre- to Post-Intervention, on average 3 hours
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 10 | 10
change in score on a scale | 2.8 (0.2) | 0.9 (0.01)

2. Other Pre Specified Outcome: Standing Duration
Description: Participants were asked to stand for as long as they could. Their standing duration was video recorded and timed in seconds. The measure reported is the change in standing time from before to after the rTMS intervention, where a positive value indicates an improvement in standing duration, a negative value indicates a worsening of standing duration, and 0 indicates no change.
Time Frame: Pre- to Post-Intervention, on average 3 hours apart
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Real rTMS Stimulation: Participants first received 900 pulse of real rTMS
- Sham rTMS Stimulation: Participants first received 900 pulse of sham rTMS
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 10 | 10
seconds | 126 (82.2) | -6.7 (29.3)

3. Other Pre Specified Outcome: Timed "Up & Go" Test (TUG) Test
Description: The TUG is a mobility test that is used to measure the basic mobility skills and gait speed of people who have neurological conditions. It includes a sit-to-stand component as well as walking 3 m, turning, and returning to the chair. People perform these tasks using regular footwear and customary walking aids. The measured outcome is the time in seconds to complete the entire sequence. For the outcome assessment the test will be videotaped and scored by a blind rater. We calculated the change between two time points (pre intervention value minus post intervention value)
Time Frame: Pre- to Post-Intervention
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Real rTMS Stimulation: rTMS will be delivered over each cerebellar hemisphere, using a 70mm figure-of-eight coil connected to a Magstim RapidStim2 machine while positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere.
  Magstim RapidStim2: Application of repetitious transcranial magnetic stimulation (TMS) pulses using Magstim RapidStim2 to a specific brain target at predefined stimulation parameters.
  Fahn-Tolosa-Marin Tremor Rating Scale (TRS): All participants will receive a clinical assessment of tremor severity by using the TRS test.
  Timed "Up & Go" Test (TUG) test: All participants will receive a clinical assessment of basic mobility skills by using the TUG test.
  10m walk test: All participants will receive a clinical assessment of walking speed by using the walk test.
  Tremor electrophysiology: All participant tremors will by analyzed using an EMG system
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
- Sham rTMS Stimulation: Patients randomized to receive sham treatment will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using sham Magstim RapidStim2 Placebo which produces discharge noise and vibration similar to the real coil without stimulating the cerebral cortex. However, in addition to obvious coil discharge noise, rTMS also causes electrical stimulation of the scalp. The investigator will simulate this experience by attaching surface electrodes underneath the sham coil and in contact with the scalp.
  Sham Magstim RapidStim2: Same procedure as real rTMS without stimulating the cerebral cortex.
  Fahn-Tolosa-Marin Tremor Rating Scale (TRS): All participants will receive a clinical assessment of tremor severity by using the TRS test.
  Timed "Up & Go" Test (TUG) test: All participants will receive a clinical assessment of basic mobility skills by using the TUG test.
  10m walk test: All participants will receive a clinical assessment of walking speed by using the walk test.
  Tremor electrophysiology: All participant tremors will by analyzed using an EMG system
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 10 | 10
seconds | 13 (1.5) | 12 (1.6)

ADVERSE EVENTS:
Time Frame: approximately 2 weeks
Groups:
- Sham rTMS Stimulation: Patients randomized to receive sham treatment will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using sham Magstim RapidStim2 Placebo which produces discharge noise and vibration similar to the real coil without stimulating the cerebral cortex. However, in addition to obvious coil discharge noise, rTMS also causes electrical stimulation of the scalp.
  Sham Magstim RapidStim2: Same procedure as real rTMS without stimulating the cerebral cortex.
  Fahn-Tolosa-Marin Tremor Rating Scale (TRS): All participants will receive a clinical assessment of tremor severity by using the TRS test.
  Timed "Up & Go" Test (TUG) test: All participants will receive a clinical assessment of basic mobility skills by using the TUG test.
  10m walk test: All participants will receive a clinical assessment of walking speed by using the walk test.
  Tremor electrophysiology: All participant tremors will by analyzed using an EMG system
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT02441985/Prot_SAP_000.pdf